CLINICAL TRIAL: NCT04812470
Title: A Phase I Study Using Hepatic Arterial Infusion of Autologous Tumor Infiltrating Lymphocytes in Patients With Melanoma and Liver Metastases
Brief Title: Hepatic Arterial Infusion of Autologous Tumor Infiltrating Lymphocytes in Patients With Melanoma and Liver Metastases
Acronym: HAITILS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vastra Gotaland Region (Other Government)
Collaborators: Miltenyi Biomedicine GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2020-006126-31
Record Dates: First submitted 2021-03-05; First posted 2021-03-23 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Metastatic Uveal Melanoma; Metastatic Cutaneous Melanoma
Keywords: Adoptive Cell Transfer; Lymphocytes, Tumor-Infiltrating; Interleukin-2; Melphalan; Antineoplastic Agents, Immunological; Hepatic arterial infusion; bioreactor
MeSH Terms: conditions — Uveal Melanoma; Melanoma | interventions — Melphalan; Interleukin-2

STUDY DESIGN:
Intervention Model Description: dose escalation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Autologous tumor infiltrating lymphocytes (TIL) (Experimental): Autologous TIL administered via hepatic arterial infusion followed by low dose Interleukin-2 after preconditioning chemotherapy with Melphalan.
  Interventions: Drug: Autologous Tumor Infiltrating Lymphocytes; Drug: Melphalan; Drug: Interleukin-2

INTERVENTIONS:
Drug: Autologous Tumor Infiltrating Lymphocytes — Administered via hepatic arterial infusion
Drug: Melphalan — Melphalan will be administered once as an intravenous infusion.
Drug: Interleukin-2 — After TIL infusion, Interleukin-2 will be administered subcutaneously once daily for up to 14 days.

SUMMARY:
The purpose of this study is to evaluate the feasibility, safety and tolerability of treatment with autologous tumor infiltrating lymphocytes (TIL) administered via hepatic arterial infusion in patients with liver metastases (including but not restricted to) of malignant melanoma.

ELIGIBILITY:
Inclusion Criteria:

1. Patients 18-75 years of age on the day of signing informed consent.
2. Patient is willing and able to provide written informed consent and comply with study procedures. Written informed consent must be signed and dated before the start of specific protocol procedures.
3. Patient must have a histologically/cytologically confirmed diagnosis of:

   * stage IV uveal melanoma with or without any previous systemic therapy OR
   * stage IV cutaneous melanoma with confirmed progression following at least one or two prior systemic therapies including a programmed cell death protein-1 (PD-1) inhibitor with or without a CTLA-4 inhibitor; and if BRAF V600 mutation-positive, also a BRAF inhibitor or a BRAF inhibitor in combination with a MEK inhibitor.
4. Measurable disease by computed tomography (CT) per RECIST 1.1 criteria with at least one target lesion identified in the liver and where the distribution pattern of metastasis is predominantly engaging the liver as judged by the investigator.
5. At least one resectable lesion in the liver (or aggregate of lesions resected) of a minimum size of 0.5 cm in diameter post- resection to generate TILs.
6. ECOG performance status of 0 - 2.
7. Female patient of childbearing potential should have a negative urine or serum pregnancy test within 72 hours prior to receiving the first treatment. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
8. Female patients of childbearing potential must be willing to use a highly efficient method of contraception (Pearl index <1), for the course of the study through 120 days after the last dose of study medication.
9. Male patients with women of childbearing potential partners must agree to use a condom for contraception, starting with the first dose of study therapy through 120 days after the last dose of study therapy.

Exclusion Criteria:

1. Life expectancy of less than 3 months.
2. History of interstitial lung disease (ILD) or (non-infectious) pneumonitis.
3. Reduced renal function defined as S- Creatinine >=1.5xULN or Creatinine Clearance < 40 mL/min, calculated using the Cockroft and Gault formula.
4. Reduced hepatic function (defined as ASAT, ALAT, bilirubin > 3*ULN and PK- INR > 1.5) or medical history of liver cirrhosis or portal hypertension.
5. Hemoglobin <90 g/L or platelets <100x109/L or neutrophils <1.5x109/L
6. Use of live vaccines four weeks before or after the start of study.
7. History of severe hypersensitivity reactions to monoclonal antibodies.
8. Active infection.
9. Infection of human immunodeficiency virus (HIV), acquired immunodeficiency syndrome (AIDS), hepatitis B or hepatitis C.
10. Active autoimmune disease or a history of known or suspected autoimmune disease.
11. A condition requiring systemic treatment with either corticosteroids (>10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids and adrenal replacement doses >10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease.
12. Concomitant therapy with any other anti- cancer therapy, concurrent medical conditions requiring use of immunosuppressive medications or use of other investigational drugs.
13. Has a known additional malignancy of other diagnosis that is progressing or requires active treatment.
14. Pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of study drug.
15. A history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the patient's participation for the full duration of the study, or is not in the best interest of the patient to participate, in the opinion of the treating Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2023-02-06 (Actual); Primary Completion 2025-05-26 (Actual); Study Completion 2025-05-26 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of adverse events (AEs) and serious adverse events (SAEs) | 5 years from start of chemotherapy
  Adverse events are graded according to the NCI Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0

SECONDARY OUTCOMES:
Objective response rate (ORR) | 2 years from start of chemotherapy
  Defined by RECIST 1.1
Clinical benefit rate (CBR) | 18 weeks
  Defined by RECIST 1.1
Progression free survival (PFS) | 2 years
  Evaluation of progression-free survival
hepatic Progression free survival (hPFS) | 2 years
  Evaluation of hepatic progression-free survival
Duration of objective response (DOR) | 2 years
  Evaluation of duration of response
Overall Survival (OS) | 5 years
  Evaluation of overall survival
Evaluation of feasibility of an automated production of TILs | 2 years
  Defined as the proportion of patients included that receive treatment with the TIL product.

CONTACTS AND LOCATIONS:
Overall Officials: Lars Ny, Principal Investigator — Department of Oncology, Sahlgrenska University Hospital, Sweden
Locations (1):
- Department of Oncology, Sahlgrenska University Hospital, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No